CLINICAL TRIAL: NCT03053635
Title: A Phase Ib Trial of Intravesical Photodynamic Therapy in Patients With Non-muscle Invasive Bladder Cancer at High Risk of Progression Who Are Refractory to Bacillus Calmette-Guerin Therapy and Who Are Medically Unfit for/Refuse Cystectomy
Brief Title: Intravesical Photodynamic Therapy (PDT) in BCG Refractory High-Risk Non-muscle Invasive Bladder Cancer (NMIBC) Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Theralase® Technologies Inc. (Industry)
Collaborators: University Health Network, Toronto (Other); Medelis Inc. (Industry); WCCT Global (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TLD1433 Bladder Cancer PDT
Record Dates: First submitted 2017-02-06; First posted 2017-02-15 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Non-Muscle Invasive Bladder Cancer (NMIBC) Refractory to BCG
Keywords: Photodynamic Therapy; Non-muscle invasive bladder cancer (NMIBC); Urothelial carcinoma; Ta bladder cancer; T1 bladder cancer; Refractory to BCG
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms; Carcinoma, Transitional Cell | interventions — Photochemotherapy; 1-phenyl-3,3-dimethyltriazene; Therapeutics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 0.35 mg/cm^2 TLD1433 Bladder Dose (Experimental): TLD1433 infusion and photodynamic therapy treatment (PDT):
  TLD1433 is infused for 1 hour and photodynamic therapy treatment is performed after TLD1433 has been rinsed from the bladder. If treatment with the maximum recommended starting dose of 0.35mg/cm^2 does not raise significant safety concerns as determined by the safety monitoring committee, the therapeutic dose of TLD1433 (0.70mg/cm^2) will be used.
  Interventions: Drug: TLD1433 infusion and photodynamic therapy (PDT) treatment

INTERVENTIONS:
Drug: TLD1433 infusion and photodynamic therapy (PDT) treatment — TLD1433 is infused into the bladder, followed by repeated rinsing and treatment of bladder wall with photodynamic therapy (PDT).
  Other Names: PDT

SUMMARY:
This is a phase Ib, open-label, single-arm, single-center study conducted in Canada. Subjects with NMIBC (Ta, T1, and/or Tis) who are not candidates for or have refused radical cystectomy will be eligible for participation in the study. Bacillus Calmette-Guerin (BCG) intolerance or refractory disease are defined as inability to tolerate or failure to achieve a tumour-free state after at least one induction (a minimum of 5 instillations) followed by either a second induction (a minimum of 5 instillations) or at least 2 maintenance instillations. Subjects experiencing disease relapse within 12 months or less after finishing the second course of BCG therapy are also considered refractory. The study will consist of 2 phases. In the first phase, 3 subjects will receive PDT (TLC-3200 System) employing 0.35 mg/cm^2 (maximum recommended starting dose) TLD1433. If treatment with the maximum recommended starting dose does not raise significant safety concerns as determined by the safety monitoring committee, an additional 6 subjects will receive PDT with 0.70 mg/cm^2 (therapeutic dose) TLD1433.

DETAILED DESCRIPTION:
10.1 Overall Study Design and Plan: Description

This is a phase Ib, open-label, single-arm, single-center study conducted in Canada. Subjects with NMIBC (Non-muscle Invasive Bladder Cancer, Ta, T1, and/or Tis) who are not candidates for or have refused radical cystectomy will be eligible for participation in this study. BCG intolerance or refractory disease are defined as inability to tolerate or failure to achieve a tumour-free state after at least one induction (a minimum of 5 instillations) followed by either a second induction (a minimum of 5 instillations) or at least 2 maintenance instillations. Subjects experiencing disease relapse within 12 months or less after finishing the second course of BCG therapy are also considered refractory.

The study will consist of 2 phases. In the first phase, 3 subjects will receive PDT employing 0.35 mg/cm^2 (maximum recommended starting dose) TLD1433 and 90 J/cm^2 of green light delivered by TLC-3200. If treatment with the maximum recommended starting dose does not raise significant safety concerns as determined by the safety monitoring committee, an additional 6 subjects will receive PDT with 0.70 mg/cm^2 (therapeutic dose) TLD1433 and 90 J/cm^2 of green light delivered by TLC-3200.

10.2 Screening Period

Subjects will be qualified for study entry by review of inclusion and exclusion criteria during the Screening Period, which will last up to 2 weeks.

10.3 Maximum Recommended Starting Dose Treatment Phase

Three subjects will receive a single instillation of 0.35 mg/cm^2 TLD1433 followed by PDT (TLC-3200 System). If treatment with the maximum recommended starting dose doesn't raise safety concerns after 1 month of patient follow-up based on the judgment of the safety monitoring committee, the study will enroll an additional 3 subjects who will receive PDT at the maximum recommended starting dose.

10.4 Follow-Up Phase

All subjects enrolled, regardless of TLD1433 dose received, will be followed until the End of Study defined as completion of all required assessments after 6 months of follow-up or earlier due to early discontinuation or withdrawal of informed consent.

During the Follow-Up Phase, information on safety and efficacy will be collected. Assessments will be conducted at Day 7, Day 30 and monthly thereafter through Month 3, and every 3 months until End of Study.

10.6 Study Drug and PDT Administration

TLD1433 for intravesical administration is supplied as a lyophilisate for suspension in Sterile Water for Injection into the bladder and is packaged in the dark in amber borosilicate glass vials which can be stored at room temperature. Just before administration, it is reconstituted with Sterile Water for Injection to obtain the final clinical dilution.

TLD1433 will be supplied by Theralase Inc. Instillations cannot be done immediately following biopsy taken by TURBT. Investigators must wait a minimum of 7 days before dosing subjects after a TURBT/biopsy and/or until any bladder wall integrity issues have resolved. Dose/volume reductions are not allowed during this study.

Upon determination of the bladder volume (during the screening period) through a voiding diary or measuring instilled water volume, TLD1433 will be diluted to the proper concentration. On day 0 (treatment day), subjects will be asked to restrict fluid intake 12 hours before study drug instillation. Study drug must be instilled into the subject's empty bladder. Before instillation, a regular transurethral catheter should be inserted and the bladder drained. A single instillation of TLD1433 will be infused intravesically for 60 min (further TLD1433 will be instilled in case of leakage), followed by 3 washes with sterile water. Bladder will be distended using a fourth instillation of sterile water to prevent folds that prevent uniform light illumination. The laser technician worksheet must be completed during the procedure and data must be promptly transferred to the corresponding eCRF page. The optical fiber (with spherical diffuser) will be positioned in the center of the bladder with the aid of TLC-3200 and will be locked in place using an endoscope holder for continuous irradiation for the total exposure time. Exposure time will be calculated based on power (measured at the end of the optic fiber before inserting though a liquid-tight lock via catheter into the urethra) and bladder surface area to match the desired light dose at the bladder wall. Green laser light (wavelength = 532 nm, energy = 90 J/cm^2) will be irradiated using the spherical cavity diffuser.

10.6.1 Dosing Schedule

A single whole bladder intravesical PDT with TLD1433 and the TLC-3200 System is planned.

10.6.2 PDT Disruption

Only those patients in whom no papillary tumours remain after TURBT will be treated on this protocol. If one or more papillary tumours are seen at the time of cystoscopy for laser light application (maximum 6 weeks after TURBT), a patient must not be treated with the TLC-3200 System as scheduled, even though previously instilled with TLD1433. Procedures will be followed as though the tumour were first detected at the 90-day follow-up evaluation. The patient may then be treated in whatever manner the physician deems appropriate. However, such patients must be followed for collection of safety information for at least 30 days after TLD1433 instillation, even though alternate therapy may have been initiated during this time. Adverse experiences, weekly assessment of urinary symptoms, and the results of laboratory tests of blood and urine will be recorded. Full disclosure of the details of any alternate therapy or other medications given during the 30-day observation period (e.g., drug, dose, route, frequency and dates of administration) must be provided. After this 30-day period, an interim medical history will be taken and the patient will undergo a physical examination (including ECG), clinical laboratory tests, a Karnofsky Performance Status rating, and an assessment of urinary symptoms and adverse experiences. The patient will then be considered off study.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent/assent for the trial.
2. Be > 18 years of age on day of signing informed consent.
3. Have histologically confirmed NMIBC (T1, Ta, and/or Tis) according to the 2004 World Health Organization (WHO) classification within 8 weeks prior of treatment initiation. Participants with tumours of mixed transitional / non-transitional cell histology are eligible, but urothelial carcinoma must be the predominant histology. Participants with predominant or exclusively non-urothelial histology are not eligible. Confirmation of histology, grade and stage will be performed by local review and must be completed prior to enrolment.
4. For participants with Ta and T1, they must have undergone complete TURBT defined as absence of resectable disease after at least 2 cystoscopy / TURBT procedures. The most recent cystoscopy must have been performed no longer than 8 weeks prior to the first dose of trial treatment.
5. Have been considered intolerant or refractory to first-line BCG therapy defined as inability to tolerate or failure to achieve a tumour-free state after at least one induction (minimum of 5 instillations) followed by at either a second induction (minimum of 5 instillations) or at least 2 maintenance instillations. Participants experiencing disease relapse within 12 months or less after finishing the second course of BCG therapy are also considered refractory.
6. Are not candidates for cystectomy on medical grounds or refuse radical cystectomy.
7. Have a performance status of 70 or more on the Karnofsky Performance Status Scale as assessed within 28 days prior to treatment initiation.
8. Have no evidence of upper urothelial carcinoma (involving the upper urinary tract or the urethra) (confirmed by staging to exclude extravesical disease, which may include radiological imaging and/or biopsy) within 3 months of treatment initiation. If previous work up occurred more than 3 months prior to treatment initiation, staging for extravesical disease must be repeated prior to enrolment in order to determine eligibility.
9. Have satisfactory bladder function. Ability to retain instillate for a minimum of 1 hour, even with premedication.
10. Are available for the duration of the study including follow-up (approximately 12 months).
11. Female participants of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
12. Female participants of childbearing potential must be willing to use 2 methods of birth control (oral contraceptive, pills, diaphragm, or condoms) or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Participants of childbearing potential are those who have not been surgically sterilized or have not been free from menses for >1 year.

Male participants must agree to use an adequate method of contraception (oral contraceptive, pills, diaphragm, or condoms) starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

1. Past or current muscle invasive (i.e., T2, T3, T4) or metastatic urothelial carcinoma.
2. Has concurrent extravesical (i.e. urethra, ureter or renal pelvis) non-muscle invasive transitional cell carcinoma of the urothelium.
3. Have a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer. A history of prostate cancer that was treated with definitive intent (surgically or through radiation therapy) is acceptable, provided that the following criteria are met: Stage T2N0M0 or lower; Prostate-Specific Antigen undetectable for 5 years while off androgen deprivation therapy.
4. Have a known psychiatric or substance abuse disorder that would interfere with meeting the requirements of the trial.
5. Have a history or current evidence of any condition, therapy, surgery or laboratory abnormality that, in the opinion of the investigator, might confound the results of the trial, interfere with the participant's participation in the trial, or is not in the best interest of the participant to participate.
6. Currently receiving any photosensitizing medications.
7. Have a known hypersensitivity to ruthenium.
8. Currently receiving treatment with a prohibited concomitant therapy (refer to 12.2.1, Prohibited Medications).
9. Participated in a study with an investigational agent or device within 3 months from the first dose of current study treatment.
10. Prior treatment with an intravesical chemotherapeutic agent within 3months of the first dose of current study drug, with the exception of a single perioperative dose of chemotherapy immediately post-TURBT (not considered treatment).
11. Have an active infection requiring systemic therapy, including active or intractable urinary tract infection (UTI), in the last month.
12. Has any contraindication to general or spinal anesthesia.
13. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the participant's participation for the full duration of the trial, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
14. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment.
15. Known history of Human Immunodeficiency Virus (HIV) (HIV-1/2 antibodies).
16. Known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., hepatitis C virus (HCV) RNA [qualitative] is detected).
17. Received a live virus vaccine within 30 days of planned start of trial treatment.
18. Have a diagnosis of psoriasis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-12-21 (Actual); Primary Completion 2018-08-09 (Actual); Study Completion 2018-08-09 (Actual)

PRIMARY OUTCOMES:
Safety Analysis of TLD1433 and PDT assessed with the incidence and severity of Adverse Effects. | Up to the completion of follow-up phase (180 days)
  Adverse events (AE) summaries will be provided showing the number and percentage of participants who experienced at least 1 AE. These summaries will be presented by body system and preferred term. Severe AEs (SAEs) and AEs resulting in discontinuation will be summarized separately in a similar fashion.

SECONDARY OUTCOMES:
Pharmacokinetic Analysis | Blood (prior to drug, 1h, 4h, 8h, 24h, and 72h post drug). Urine (prior to drug, 8h, 24h, and 72h post drug)
  Pharmacokinetics (PK) parameters for blood and urine will be calculated using non-compartmental analysis. The Area Under the Curve (AUC0-t) will be calculated with the linear trapezoidal method.

OTHER OUTCOMES:
Exploratory Efficacy Analysis: The exploratory outcome endpoint is Recurrence-Free Survival (RFS). | The overall efficacy will be evaluated during the course of the study (at 3 and 6 months)
  RFS is defined as the interval from Day 0 to documented recurrence or death from any cause, whichever occurs first. Recurrence is defined as any new tumor growth (i.e. any biopsy-confirmed new or recurrent tumor), evaluated at 90 days for the first three patients treated at the Maximum Recommended Starting Dose (MRSD) (0.35 mg/cm2) and primarily at 90 days for the last six patients treated at the Therapeutic Dose (0.70 mg/cm2) and secondarily one hundred and eighty (180) days post treatment. For patients who are lost to follow-up or withdraw from the study before recurrence or death, the RFS will be censored at last disease assessment (i.e.: date of last biopsy or cystoscopy); for participants who start new anti- cancer treatment (i.e.: chemotherapy, immunotherapy or radiotherapy) or undergo a cystectomy, the RFS will be censored at the last disease assessment (i.e.: date of last biopsy or cystoscopy) before the start of the new anti-cancer therapy or cystectomy.

CONTACTS AND LOCATIONS:
Overall Officials: Girish Kulkarni, MD, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided